CLINICAL TRIAL: NCT04815889
Title: The PLUSS Model: a Study Protocol for Evaluation of a Multi-professional and Intersectoral Working Model to Detect Neurodevelopmental Difficulties in Preschool Children as Well as to Provide Parental Support
Brief Title: Early Detection and Intervention in Developmental Delay / Behavioral Problems in Preschool Children - PLUSS
Acronym: PLUSS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Jönköping County (Other Government)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Screening
Other Study IDs: RJonkopingC
Record Dates: First submitted 2021-03-16; First posted 2021-03-25 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Developmental Delay; Behavioural Problem; Neurodevelopmental Delay
Keywords: Behavioural problems; Developmental Delay; Intervention; Preschool children; Screening
MeSH Terms: conditions — Learning Disabilities; Mental Disorders | interventions — Schools, Nursery

STUDY DESIGN:
Intervention Model Description: All families receive the first interventions, which are PRIMUS parent education and teacher education. Then the families receive different interventions based on need. The control group receives treatment as usual.
Who Masked: Participant
Masking Description: Children who are referred to a Child Health psychologist at the age of 1.5-4 (mostly after 2.5 years of supervision at the Child Health Nurse).
  Informants are parents, preschool teachers, child health care psychologists and nurses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Recruitment of the control group is done through the county parts that have not yet been included in the clinical trial of new methods. This means that children / families are not withheld from treatment they would otherwise receive.
- PRIMUS parent training group and preschool teacher training group (Active Comparator): The parents have undergone PRIMUS Group-based parent support program for 5 half days This parenting education for preschool children with developmental problems but without the requirement of diagnosis Hellström (2019) has been designed and tested in other parts of the country but not scientifically validated, which can be done in this study. The preschool teachers may participate for half a day in education together with the parents as a practical implementation in the child's everyday life.
  Interventions: Behavioral: PRIMUS parent training Group
- Demand-driven intervention (Other): The PLUSS toddler team makes a "management plan" as referral to Habilitation Center, Child and Adolescent Psychiatry, Speech Therapist, or interventions eg:
  * Support in the child's everyday environment home / preschool
  * Targeted parent training group: toilet, sleep, food, everyday structure, handle behavioural problems
  * Web Courses Each individual intervention is evaluated afterwards with the study questionnaire.
  Interventions: Behavioral: PRIMUS parent training Group

INTERVENTIONS:
Behavioral: PRIMUS parent training Group — The parents offered a PRIMUS Group-based parent support program for 5 half days. This parenting education for preschool children with developmental problems but without the requirement of diagnosis Hellström (2019) has been designed and tested in other parts of the country but not scientifically validated, which can be done in this study. The teachers will be offered a teacher group for half a day together with the parents.
  For those families who need more intervention the PLUSS toddler team (from the specialist Healthcare) is established.
  The PLUSS toddler team makes a "management plan" as referral to Habilitation Center, Child and Adolescent Psychiatry, Speech Therapist, or interventions eg:
  * Support in the child's everyday environment home / preschool
  * Targeted Parent Groups: toilet, sleep, food, everyday structure, handle behavioural problems
  * Web courses
  Other Names: Preschool and teacher training Group; Emotional Regulation parentgroup; Individual efforts in preschool; Individual efforts to parents
  Arms: Demand-driven intervention; PRIMUS parent training group and preschool teacher training group

SUMMARY:
The PLUSS (Mental health, learning, development, collaboration around preschool children) is a collaborative project involving guardians, Jönköping County´s health care, preschools and social services. The project studies the implementation of a "One way in"-model that provides coordinated services to screen, evaluate and treat toddlers with behavioral problems. The project also provides parental interventions and education for preschool teachers.

The study aims to investigate a) implementation of the PLUSS model, b) effectiveness of the model and the included parental training program on behavioral problem and their longitudinal development among preschool children, c) parental wellbeing and satisfaction. In the long term, the goal is to reduce mental health problems among children, adolescents and their families and to provide support for a functioning everyday life.

DETAILED DESCRIPTION:
The Jönköping Health Care managers for Child Health Care, Habilitation Center, Child and Adolescent Psychiatry and Rehabilitation Center (Speech Therapist) searched at 2018 government funding during this collaborative PLUSS-project. They have since money was awarded to the project in 2019, been formatted as a steering group for these clinical research project. An operational interprofessional working group appointed by the managers to conduct clinical and research work under the guidance of a disputed project manager of 40%. Information about the PLUSS-project and collaboration with the municipalities' activities (preschool and social services) started in 2019.

Ethics approval has been granted by the National Ethics Board (#2019-04839). Informed consent is obtained from all actors: both parents, managers, preschool educators, CHP and CHN. All data is registered with fp-number and is encoded directly at the time of collection considering the protection of privacy. Code template for translation between fp-no and the test subject can be found in a logbook that is kept inaccessible to unauthorized persons. The results are reported only at the group level, where no personal data will be recognizable. All data processing takes place following Swedish data law. The parents have been informed that they receive the same care whether they participate in the study or not. The project could cause concern for the parents as they answer the questionnaire and become aware of the child's possible problem. Here it is an advantage that the CHP uses the questionnaire in the assessment interview so that the parent has the opportunity to ask questions or talk about his child's needs and strengths. Recruitment of the control group is done through the county parts that have not yet been included in the clinical trial of new methods. This means that children/families are not withheld from treatment they would otherwise receive.

After the assessment interview and with the parents' consent, the Child Health psychologist contacts the child's preschool. The preschool manager and preschool teacher may consent to participate in the study and the preschool teacher answers questionnaires. The behavior of the children in the preschool will be paid extra attention to the teachers as they are asked to assess the behavior of the individual child. This could lead to children's problem behavior being highlighted in a way that can change how teacher's behaved towards individual children. However, an exaggerated emphasis on the negative is counteracted by the teacher being also asked to estimate the child's mental health in the form of commitment and social interaction. The project focuses on efforts in the child's environment that are helpful to all children, not just those with special needs.

ELIGIBILITY:
Inclusion Criteria:

* Development Delay
* Interaction, contact difficulties
* Language and communication difficulties
* Difficulties in everyday function
* Motor difficulties
* Concentration / hyperactive
* Self-regulation
* Acting / boundaries
* Anxiety
* No claim to diagnosis

Exclusion Criteria:

* Not only support in the parent role, without any of the problems above.

Ages: 18 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Strengths and Difficulties questionnaire (SDQ | Change from baseline, pre intervention.Up to 24 weeks.
  Measured with Behavioral problems with 25 items divided into 5 subscales of 5 items each, generating scores for 4 problem subscales: Conduct problems, Hyperactivity, Emotional problems and Peer problems, and 1 strength subscale: Prosocial behaviours. Responses are given on a 3-point Likert scale: (0) "not true" (1) "somewhat true" (2) "certainly true". The total scores for the behavioural difficulties scale are maximum 50 points (worse outcome), minimum 0 points (best outcome).
  The impairment supplement questions, which describe how behavioural problems affect the child's level of functioning, are subsequently included in the impact score. Ratings for these 8 impairment supplement questions are: (0) "not at all" and (0) "only a little" (1) "quite a lot" and (2) "a great deal". Maximum 16 points (worse outcome), minimum 0 points (best outcome) (Goodman, 2016). SDQ is validated and proposed cut-offs are available for Swedish conditions (Goodman, 2016; Gustafsson et al, 2016).

SECONDARY OUTCOMES:
Children's engagement questionnaire (CEQ) | Change from baseline, pre intervention. Up to 24 weeks.
  Functioning, Mental Health: Children's engagement questionnaire (CEQ) is a form of 29 questions. Compared with the following alternatives: (1) almost never happens (2) sometimes happens (3) happens quite often or (4) happens very often. The maximum score is 116 and the minimum score is 0. It is positive to have as high a score as possible. It measures children's targeted engagement and social interaction in preschool children's everyday life and is validated for Swedish conditions (Mc William, 1991).
Measured with the Observation instrument Joint Attentment observations (JA-OBS) | Baseline when the child is on a 2.5 year check-up with the CHC nurse
  Autism spectrum: Measured with the Observation instrument Joint Attentment observations (JA-OBS) how includes 5 questions and are a Autism spectrum screening instrument (Sweden County Councils and Regions, 2018). Maximum score = 5, minimum score = 0. 4-5 points show no signs of autism spectrum symptoms.
Psychosocial problems in the family (LAPS) | Change from baselaine, pre intervention. Up to 24 weeks.
  Psychosocial problems in the family: LAPS, translated from Finnish where this form is filled in by Health Care staff. The form has been developed and tested within the framework of the project for the development of mental health work among children 2007-2009 (Mäki et al, 2014). LAPS consists of 16 items with 3 answer options. The instrument is not validated or standardized for Swedish conditions. There are cut-off figures based on Finnish conditions that show when support for the family should be offered (5-7 points for primary care and over 8 points for specialist care). The form is filled in by the BHV psychologist at the first assessment interview with the guardians. To be filled in by the BHV psychologist and can be graded in no (0), mild (1) and severe symptoms (2). The maximum score on the instrument is 32 and then indicates severe symptoms in all items.

CONTACTS AND LOCATIONS:
Overall Officials: Berit M Gustafsson, PhD, Principal Investigator — Region Jönköping County "RJonkopingC"
Locations (1):
- Region Jönköping County "RJonkopingC", Eksjö, Jönköping County, Sweden

IPD SHARING:
Plan to Share IPD: No
We are not supposed to share the data of the ethical considerations.

REFERENCES:
- [Result] Gustafsson BM, Korhonen L. A Multiprofessional and Intersectoral Working Model to Detect and Support Preschool Children With Neurodevelopmental Difficulties (PLUSS Model): Protocol for an Evaluation Study. JMIR Res Protoc. 2022 Jun 15;11(6):e34969. doi: 10.2196/34969. PMID 35704376
- [Derived] Gustafsson BM, Steinwall S, Korhonen L. Multi-professional and multi-agency model PLUSS to facilitate early detection and support of pre-school children with neurodevelopmental difficulties - a model description. BMC Health Serv Res. 2022 Mar 30;22(1):419. doi: 10.1186/s12913-022-07815-8. PMID 35354442
- See also: A Multiprofessional and Intersectoral Working Model to Detect and Support Preschool Children With Neurodevelopmental Difficulties (PLUSS Model): Protocol for an Evaluation Study — https://pubmed.ncbi.nlm.nih.gov/35704376/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35704376/
- Available data/document: Study Protocol — https://pubmed.ncbi.nlm.nih.gov/35704376/